CLINICAL TRIAL: NCT04011215
Title: Determining Effects of Superfine Sheep Wool in INfantile Eczema (DESSINE 2): a Multicentre Randomized Crossover Study
Brief Title: Wool Clothing for the Management of Childhood Atopic Dermatitis (DESSINE2)
Acronym: DESSINE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Australian Wool Innovation Ltd (Unknown); Northwestern University (Other); United Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019.034
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- wool-first (wool X standard) (Experimental): superfine merino wool clothing to be worn for 6 weeks followed by 6 weeks of standard clothing
  Interventions: Other: wool clothing; Other: standard clothing
- standard-first (standard X wool) (Active Comparator): standard clothing to be worn for 6 weeks followed by 6 weeks of superfine merino wool clothing
  Interventions: Other: wool clothing; Other: standard clothing

INTERVENTIONS:
Other: wool clothing — superfine merino wool ensembles for baby/child wear
Other: standard clothing — Standard clothing refers to the clothing normally worn by the infant/child. This will not be superfine merino wool as superfine merino is not generally available for baby wear. The exact nature of the standard clothing will be recorded by investigators. From previous data we expect it to be primarily cotton.

SUMMARY:
The study is a sequentially recruited, cross-over-cohort, outpatient-based evaluation of the effectiveness of wool clothing, as compared to standard clothing, in reducing the severity of childhood atopic dermatitis (eczema) over two consecutive six-week periods.

DETAILED DESCRIPTION:
The study will aim for a sample size of approximately 150 participants (equally distributed between 3 international sites) between the ages of 3 months and 5 years referred to the respective Dermatology Departments for management of moderate to severe atopic dermatitis. They will be sequentially recruited and randomized to the wool-to-standard clothing arm or standard clothing-to-wool arm.

The study will run for 12 weeks for each participant with two consecutive 6-week periods for each intervention, either of wool followed by standard clothing or standard followed by wool clothing. Participants will be assessed by a blinded trained researcher, at their initial appointment, 3 weeks, 6 weeks, 9 weeks and 12 weeks post commencement of the first intervention.

The primary outcome is the severity of atopic dermatitis at 6 weeks post commencement of each intervention i.e.at week 6 and week 12. Severity of atopic eczema will be measured using the Eczema Area and Severity Index (EASI).

Secondary outcomes include the severity and change in the severity of eczema using the EASI at 3 weeks, the validated Investigators Global Assessment for atopic dermatitis (vIGA-AD™) score and quality of life assessment using the children's Dermatology Life Quality Index (cDLQI) at 3 and 6 weeks of each 6 week intervention period, as well as weekly Patient Oriented SCORing Atopic Dermatitis index (PO-SCORAD) scores.

ELIGIBILITY:
Inclusion Criteria:

* Is aged between 3 months and 5 years of age at the time of recruitment
* Has moderate to severe eczema as determined by an EASI score of 7 or above at their initial visit
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participants behalf

Exclusion Criteria:

* Has a known allergic contact dermatitis to wool or merino wool
* Is unable to attend all scheduled visits
* Has unstable eczema defined by an escalation of treatment requirements during the preceding 6 weeks. This would include flares of AD for any reason including infection, food allergy etc.
* Use of systemic corticosteroids within 6 weeks of study start.
* Any medical reason that is considered by the principal investigator to preclude enrolment.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | week 3 of each 6 week period (ie week 6 and 12)
  blinded assessor administered EASI (units on a scale), will assess change from baseline. A score is obtained ranging from 0-72 based on erythema, papulation, excoriation and lichenification, each graded 0-3 for each of four body regions (head and neck, upper limbs, trunk, lower limbs) that are weighted according to surface area representation. A higher number indicates increased severity.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | week 3 of each 6 week period (ie week 3 and 9)
  blinded assessor administered EASI (units on a scale), will assess change from baseline.
validated Investigators Global Assessment for atopic dermatitis (vIGA-AD™) score | week 3, 6, 9, 12
  blinded assessor administered vIGA-AD™ score (units on a scale), will assess change from baseline. This score assesses erythema, induration/papulation, lichenification and oozing/crusting on ascale of 0 to 4. A high score reflects greater severity.
children's Dermatology Life Quality Index (cDLQI) | week 3, 6, 9, 12
  patient administered cDLQI questionnaire (units on a scale), will assess change from baseline. Ten questions are each scored from 0 to 3, the total score ranging from 0-30. A higher score reflects greater impairment of quality of life.
Patient Oriented SCORing Atopic Dermatitis score (PO-SCORAD) | weekly over 12 weeks
  patient completed PO-SCORAD score (units on a scale). It measures global severity using a scale ranging from 0 to 103, based on disease extent, six morphological parameters and two subjective markers (itch and sleep disturbance). High scores reflect greater severity.
Topical medication use | daily over 12 weeks
  questionnaire (number of times per day medication is applied; the name and strength of medication will be noted). This will be compared with baseline use.
Topical moisturiser use | weekly over 12 weeks
  questionnaire to determine number of times per day moisturiser is applied. This will be compared with baseline use.

CONTACTS AND LOCATIONS:
Overall Officials: John C Su, FACD, FRACP, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Northwestern University, Skin Disease Research Center, Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the DESSINE2 trial will be available six months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing john.su@mcri.edu.au
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication of the primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the DESSINE2 Trial Steering Committee must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.

REFERENCES:
- [Background] Su JC, Dailey R, Zallmann M, Leins E, Taresch L, Donath S, Heah SS, Lowe AJ. Determining Effects of Superfine Sheep wool in INfantile Eczema (DESSINE): a randomized paediatric crossover study. Br J Dermatol. 2017 Jul;177(1):125-133. doi: 10.1111/bjd.15376. Epub 2017 Jun 12. PMID 28182252